CLINICAL TRIAL: NCT03859323
Title: A Randomized, Double-blind, Placebo-controlled, Phase 1 Study to Assess the Safety, Tolerability, and Pharmacokinetics of Ascending, Subcutaneous, Single and Multiple Doses of SHP681 (GLP-2 Analog-Fc Fusion) in Healthy Adult Subjects
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of Ascending, Subcutaneous, Single and Multiple Doses of SHP681 (Glucagon-like Peptide-2 [GLP-2] Analog-Fc Fusion) in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SHP681-101
Record Dates: First submitted 2019-02-28; First posted 2019-03-01 (Actual); Results first posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Single Ascending Dose (SAD): 0.2 mg/kg (Experimental): Participants will receive single subcutaneous (SC) injection of 0.2 mg/kg SHP681 in the abdomen.
  Interventions: Drug: SHP681
- Single Ascending Dose (SAD): 0.5 mg/kg (Experimental): Participants will receive single SC injection of 0.5 mg/kg SHP681 in the abdomen.
  Interventions: Drug: SHP681
- Single Ascending Dose (SAD): 1 mg/kg (Experimental): Participants will receive single SC injection of 1 mg/kg SHP681 in the abdomen.
  Interventions: Drug: SHP681
- Single Ascending Dose (SAD): 2 mg/kg (Experimental): Participants will receive single SC injection of 2 mg/kg SHP681 in the abdomen.
  Interventions: Drug: SHP681
- Single Ascending Dose (SAD): 4 mg/kg (Experimental): Participants will receive single SC injection of 4 mg/kg SHP681 in the abdomen.
  Interventions: Drug: SHP681
- Single Ascending Dose (SAD): Placebo (Placebo Comparator): Participants will receive single SC injection of placebo matched to SHP681 in the abdomen.
  Interventions: Other: Placebo
- Multiple Ascending Dose (MAD): 0.2 mg/kg (Experimental): Participants will receive SC injection of 0.2 mg/kg SHP681 once weekly for 5 weeks in the abdomen.
  Interventions: Drug: SHP681
- Multiple Ascending Dose (MAD): 0.5 mg/kg (Experimental): Participants will receive SC injection of 0.5 mg/kg SHP681 once weekly for 5 weeks in the abdomen.
  Interventions: Drug: SHP681
- Multiple Ascending Dose (MAD): 1 mg/kg (Experimental): Participants will receive SC injection of 1 mg/kg SHP681 once weekly for 5 weeks in the abdomen.
  Interventions: Drug: SHP681
- Multiple Ascending Dose (MAD): 2 mg/kg (Experimental): Participants will receive SC injection of 2 mg/kg SHP681 once weekly for 5 weeks in the abdomen.
  Interventions: Drug: SHP681
- Multiple Ascending Dose (MAD): 4 mg/kg (Experimental): Participants will receive SC injection of 4 mg/kg SHP681 once weekly for 5 weeks in the abdomen.
  Interventions: Drug: SHP681
- Multiple Ascending Dose (MAD): Placebo (Placebo Comparator): Participants will receive SC injection of placebo matched to SHP681 once weekly for 5 weeks in the abdomen.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SHP681 — Participants will receive SC injection of SHP681 in the abdomen.
  Arms: Multiple Ascending Dose (MAD): 0.2 mg/kg; Multiple Ascending Dose (MAD): 0.5 mg/kg; Multiple Ascending Dose (MAD): 1 mg/kg; Multiple Ascending Dose (MAD): 2 mg/kg; Multiple Ascending Dose (MAD): 4 mg/kg; Single Ascending Dose (SAD): 0.2 mg/kg; Single Ascending Dose (SAD): 0.5 mg/kg; Single Ascending Dose (SAD): 1 mg/kg; Single Ascending Dose (SAD): 2 mg/kg; Single Ascending Dose (SAD): 4 mg/kg
Other: Placebo — Participants will receive SC injection of placebo matched to SHP681 in the abdomen.
  Arms: Multiple Ascending Dose (MAD): Placebo; Single Ascending Dose (SAD): Placebo

SUMMARY:
The purpose of the study is to assess the safety and tolerability of single and multiple ascending subcutaneous (SC) doses of SHP681 in healthy adult participants.

DETAILED DESCRIPTION:
The study consists of a single ascending dose (SAD) portion and a multiple ascending dose (MAD) portion.

The study duration for the SAD portion of the study consists of a screening period of up to 28 days and 1 treatment period of 29 days. SAD portion of the study contains 5 cohorts and dose escalation will proceed sequentially to assess the following single SC doses of SHP681 or SHP681 matched placebo: 0.2 milligram per kilogram (mg/kg), 0.5 mg/kg, 1 mg/kg, 2 mg/kg, and 4 mg/kg.

The study duration of the MAD portion comprises of a screening period up to 28 days and a treatment period of 57 days for each cohort. MAD portion of the study contains 6 cohorts and dose escalation will proceed sequentially to assess the following SC doses of SHP681 or SHP681 matched placebo: 0.2 mg/kg, 0.5 mg/kg, 1 mg/kg, 2 mg/kg, and 4 mg/kg once weekly for 5 weeks till 5 cohorts and the 6th cohort will receive 4 mg/kg SHP681 or matched placebo every 2 weeks over a 6-week period (3 doses).

ELIGIBILITY:
Inclusion Criteria:

* Ability to voluntarily provide written, signed, and dated informed consent to participate in the study.
* An understanding, ability, and willingness to fully comply with study procedures and restrictions.
* Age 18-50 inclusive at the time of consent. The date of signature of the informed consent is defined as the beginning of the screening period. This inclusion criterion will only be assessed at the first screening visit.
* Male, or non-pregnant, non-lactating female who agrees to comply with any applicable contraceptive requirements of the protocol or females of non-childbearing potential.
* Considered "healthy" by the investigator. Healthy status is defined by absence of evidence of any active or chronic disease or condition based on a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead electrocardiogram (ECG), hematology, blood chemistry, and urinalysis.
* Body mass index between 18.0 kilograms per square meter (kg/m^2) and 30.0 kg/m^2 inclusive with a body weight 50-100 kg (110-220 pounds [lbs]). This inclusion criterion will only be assessed at the first screening visit.

Exclusion Criteria:

* History of any hematological, hepatic, respiratory, cardiovascular, renal, neurological or psychiatric disease, gall bladder removal, or current or recurrent disease that could affect the action, absorption, or disposition of the investigational product, or clinical or laboratory assessments.
* Current or relevant history of physical or psychiatric illness, any medical disorder that may require treatment or render the participant unlikely to fully complete the study, or any condition that presents undue risk from the investigational product or procedures.
* Known or suspected intolerance or hypersensitivity to the investigational product(s), closely-related compounds, or any of the stated ingredients.
* Significant illness, as judged by the investigator, within 2 weeks of the first dose of investigational product.
* Known history of alcohol or other substance abuse within the last year.
* Donation of blood or blood products (example [eg], plasma or platelets) within 60 days prior to receiving the first dose of investigational product.
* Within 30 days prior to the first dose of investigational product:

  1. Have used an investigational product (if elimination half-life is less than (<) 6 days, otherwise 5 half-lives).
  2. Have been enrolled in a clinical study.
  3. Have had any substantial changes in eating habits, as assessed by the investigator.
* Use of dipeptidyl peptidase (DPP)-4 inhibitors within 30 days or 5 half-lives, whichever is greater, prior to administration of the investigational product.
* Confirmed systolic blood pressure greater than (>) 139 millimeters of mercury (mmHg) or <89mmHg, and diastolic blood pressure > 89mmHg or <49 mmHg.
* Twelve-lead ECG demonstrating corrected QT interval by Fredericia (QTcF) >450 millisecond (msec) at screening. If QTcF exceeds 450 msec, the ECG should be repeated 2 more times and the average of the 3 QTcF values should be used to determine the participant's eligibility.
* Positive screen for alcohol or illicit drugs at screening or Day -1.
* Male participants who consume more than 21 units of alcohol per week or 3 units per day. Female participants who consume more than 14 units of alcohol per week or 2 units per day.

  (1 alcohol unit equal to [=] 1 beer or 1 wine (5 ounce [oz] per 150 milliliter [mL]) or 1 liquor (1.5 oz/40 mL) or 0.75 oz alcohol).
* Positive human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody screen.
* Use of tobacco in any form (eg, smoking or chewing) or other nicotine-containing products in any form (eg, gum, patch). Ex-users must report that they have stopped using tobacco for at least 30 days prior to receiving the first dose of investigational product.
* Routine consumption of more than 2 units of caffeine per day or participants who experience headaches associated with caffeine withdrawal. (1 caffeine unit is contained in the following items: one 6 oz (180 mL) cup of coffee, two 12 oz (360 mL) cans of cola, one 12 oz cup of tea, three 1 oz (85 g) chocolate bars. Decaffeinated coffee, tea, or cola are not considered to contain caffeine).
* Prior screen failure (unless Sponsor approval is given), randomization, participation, or enrollment in this study or prior exposure to any GLP-2 analogs.
* Unresected gastrointestinal (GI) polyp, known polyposis condition, or premalignant changes in the GI tract.
* Any history of malignancy in the GI tract or treatment for any other malignancy in the previous 5 years.
* Current use of any medication (including over-the-counter, herbal, or homeopathic preparations; with the exception of hormonal replacement therapy or hormonal contraceptives and occasional use of ibuprofen or acetaminophen and pre-approved medication for sedation or other medications required during or after the endoscopy). Current use is defined as use within 14 days of the first dose of investigational product.
* Findings of subclinical hepatobiliary disease, such as gallstones, on abdominal ultrasound at screening as determined by the Investigator in consultation with the Medical Monitor.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (1):
- New Orleans Center for Clinical Research, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at single site in United States of America from 25 March 2019 (first participant first visit) and 06 January 2020 (last participant last visit).
Pre-assignment Details: This study consisted of 2 parts: Part A - single ascending dose (SAD) and Part B - multiple ascending dose (MAD). A total of 104 participants were randomized in 2 parts with 30 participants to SAD and 74 participants to MAD, out of which 95 participants completed the study.
Groups:
- Part 1: Single Ascending Dose (SAD): Placebo: Participants received single subcutaneous (SC) injection of placebo matched to SHP681 in the abdomen on Day 1.
- Part 1: Single Ascending Dose (SAD): 0.2 mg/kg: Participants received single SC injection of 0.2 milligrams per kilogram (mg/kg) SHP681 in the abdomen on Day 1.
- Part 1: Single Ascending Dose (SAD): 0.5 mg/kg: Participants received single SC injection of 0.5 mg/kg SHP681 in the abdomen on Day 1.
- Part 1: Single Ascending Dose (SAD): 1 mg/kg: Participants received single SC injection of 1 mg/kg SHP681 in the abdomen on Day 1.
- Part 1: Single Ascending Dose (SAD): 2 mg/kg: Participants received single SC injection of 2 mg/kg SHP681 in the abdomen on Day 1.
- Part 1: Single Ascending Dose (SAD): 4 mg/kg: Participants received single SC injection of 4 mg/kg SHP681 in the abdomen on Day 1.
- Part 2: Multiple Ascending Dose (MAD): Placebo: Participants received SC injection of placebo matched to SHP681 once weekly for 5 weeks in the abdomen up to Day 29.
- Part 2: Multiple Ascending Dose (MAD): 0.2 mg/kg: Participants received SC injection of 0.2 mg/kg SHP681 once weekly for 5 weeks in the abdomen up to Day 29.
- Part 2: Multiple Ascending Dose (MAD): 0.5 mg/kg: Participants received SC injection of 0.5 mg/kg SHP681 once weekly for 5 weeks in the abdomen up to Day 29.
- Part 2: Multiple Ascending Dose (MAD): 1 mg/kg: Participants received SC injection of 1 mg/kg SHP681 once weekly for 5 weeks in the abdomen up to Day 29.
- Part 2: Multiple Ascending Dose (MAD): 2 mg/kg: Participants received SC injection of 2 mg/kg SHP681 once weekly for 5 weeks in the abdomen up to Day 29.
- Part 2: Multiple Ascending Dose (MAD): 4 mg/kg: Participants received SC injection of 4 mg/kg SHP681 once weekly for 5 weeks in the abdomen up to Day 29.
- Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (Q2W): Participants received SC injection of placebo matched to SHP681 twice weekly (Q2W) for 5 weeks in the abdomen up to Day 29.
Period: Overall Study
Arm/Group | Part 1: Single Ascending Dose (SAD): Placebo | Part 1: Single Ascending Dose (SAD): 0.2 mg/kg | Part 1: Single Ascending Dose (SAD): 0.5 mg/kg | Part 1: Single Ascending Dose (SAD): 1 mg/kg | Part 1: Single Ascending Dose (SAD): 2 mg/kg | Part 1: Single Ascending Dose (SAD): 4 mg/kg | Part 2: Multiple Ascending Dose (MAD): Placebo | Part 2: Multiple Ascending Dose (MAD): 0.2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 0.5 mg/kg | Part 2: Multiple Ascending Dose (MAD): 1 mg/kg | Part 2: Multiple Ascending Dose (MAD): 2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (Q2W)
Started | 5 | 5 | 5 | 5 | 5 | 5 | 12 | 10 | 10 | 10 | 10 | 12 | 10
Completed | 5 | 5 | 4 | 5 | 5 | 4 | 11 | 10 | 10 | 8 | 9 | 10 | 9
Not Completed | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) included participants who had received at least one dose of TAK-681 or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Single Ascending Dose (SAD): Placebo | Part 1: Single Ascending Dose (SAD): 0.2 mg/kg | Part 1: Single Ascending Dose (SAD): 0.5 mg/kg | Part 1: Single Ascending Dose (SAD): 1 mg/kg | Part 1: Single Ascending Dose (SAD): 2 mg/kg | Part 1: Single Ascending Dose (SAD): 4 mg/kg | Part 2: Multiple Ascending Dose (MAD): Placebo | Part 2: Multiple Ascending Dose (MAD): 0.2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 0.5 mg/kg | Part 2: Multiple Ascending Dose (MAD): 1 mg/kg | Part 2: Multiple Ascending Dose (MAD): 2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (Q2W) | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 12 | 10 | 10 | 10 | 10 | 12 | 10 | 104
Age, Continuous [Median (Standard Deviation); unit: Years] | 33.6 (12.93) | 28.8 (7.60) | 38.0 (9.19) | 41.4 (8.32) | 33.0 (7.35) | 29.8 (3.96) | 31.2 (9.34) | 32.1 (8.63) | 32.5 (9.47) | 28.4 (9.52) | 32.7 (9.38) | 29.8 (10.38) | 32.0 (8.45) | 32.0 (9.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 3 | 0 | 2 | 3 | 1 | 3 | 6 | 2 | 5 | 2 | 33
  Male | 3 | 3 | 3 | 2 | 5 | 3 | 9 | 9 | 7 | 4 | 8 | 7 | 8 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 3 | 1 | 1 | 10
  Not Hispanic or Latino | 5 | 5 | 5 | 5 | 5 | 4 | 11 | 9 | 10 | 8 | 7 | 11 | 9 | 94
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 1 | 1 | 1 | 2 | 4 | 1 | 3 | 4 | 0 | 2 | 1 | 24
  White | 3 | 3 | 4 | 4 | 4 | 3 | 7 | 7 | 7 | 6 | 10 | 8 | 9 | 75
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious TEAEs and TEAEs Based on Severity to SHP681 in Single Ascending Dose (SAD)
Description: Adverse event (AE) was any unfavorable and unintended sign, symptom, or disease temporally associated with study or use of investigational drug product (IP), whether or not the AE was considered related to IP. TEAEs: AEs occurring or worsening at or after first dose of IP or ongoing at time of enrollment. SAE :untoward medical occurrence that at any dose met one, more of the following criteria: results in death, life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent, significant disability/incapacity, a congenital abnormality/birth defect, an important medical event. Severity: Mild: event that does not generally interfere with usual activities of daily living; Moderate: event that interferes with usual activities of daily living, causing discomfort, permanent risk of harm; Severe: AE that interrupts usual activities of daily living, significantly affects clinical status, or may require intensive therapeutic intervention.
Time Frame: From start of study drug administration up to follow-up (Day 29 for SAD)
Population: SAS included participants who had received at least 1 dose of SHP681 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Single Ascending Dose (SAD): Placebo | Part 1: Single Ascending Dose (SAD): 0.2 mg/kg | Part 1: Single Ascending Dose (SAD): 0.5 mg/kg | Part 1: Single Ascending Dose (SAD): 1 mg/kg | Part 1: Single Ascending Dose (SAD): 2 mg/kg | Part 1: Single Ascending Dose (SAD): 4 mg/kg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
Participants
  Participants with TEAEs | 3 | 3 | 2 | 4 | 3 | 2
  Participants with Serious TEAEs | 0 | 0 | 0 | 0 | 0 | 0
  Participants with Mild TEAEs | 3 | 3 | 2 | 4 | 3 | 2
  Participants with Moderate TEAEs | 0 | 0 | 0 | 0 | 0 | 0
  Participants with Severe TEAEs | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious TEAEs and TEAEs Based on Severity to SHP681 in Multiple Ascending Dose (MAD)
Description: AE was any unfavorable and unintended sign, symptom, or disease temporally associated with study or use of investigational drug product (IP), whether or not the AE was considered related to IP. TEAEs: AEs occurring or worsening at or after first dose of IP or ongoing at time of enrollment. SAE :untoward medical occurrence that at any dose met one, more of the following criteria: results in death, life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent, significant disability/incapacity, a congenital abnormality/birth defect, an important medical event. Severity: Mild: event that does not generally interfere with usual activities of daily living; Moderate: event that interferes with usual activities of daily living, causing discomfort, permanent risk of harm; Severe: AE that interrupts usual activities of daily living, significantly affects clinical status, or may require intensive therapeutic intervention.
Time Frame: From start of study drug administration up to follow-up (Day 57 for MAD)
Population: SAS included participants who had received at least 1 dose of SHP681 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Multiple Ascending Dose (MAD): Placebo | Part 2: Multiple Ascending Dose (MAD): 0.2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 0.5 mg/kg | Part 2: Multiple Ascending Dose (MAD): 1 mg/kg | Part 2: Multiple Ascending Dose (MAD): 2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (Q2W)
Number analyzed (Participants) | 12 | 10 | 10 | 10 | 10 | 12 | 10
Participants
  Participants with TEAEs | 9 | 8 | 3 | 6 | 5 | 9 | 8
  Participants with Serious TEAEs | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Participants with Mild TEAEs | 9 | 8 | 3 | 6 | 5 | 9 | 8
  Participants with Moderate TEAEs | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Participants with Severe TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Anti-drug Antibody (ADA) to SHP681 in Single Ascending Dose (SAD) at Day 29
Description: Antibody testing was conducted using an electro chemiluminescent signal method. Number of participants with ADA to SHP681 in SAD at Day 29 were reported.
Time Frame: Day 29
Population: SAS included participants who had received at least 1 dose of SHP681 or placebo. Here, the number of participants analyzed refer to the participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Single Ascending Dose (SAD): Placebo | Part 1: Single Ascending Dose (SAD): 0.2 mg/kg | Part 1: Single Ascending Dose (SAD): 0.5 mg/kg | Part 1: Single Ascending Dose (SAD): 1 mg/kg | Part 1: Single Ascending Dose (SAD): 2 mg/kg | Part 1: Single Ascending Dose (SAD): 4 mg/kg
Number analyzed (Participants) | 5 | 5 | 4 | 5 | 5 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Anti-drug Antibody (ADA) to SHP681 in Multiple Ascending Dose (MAD) at Day 36
Description: Antibody testing was conducted using an electro chemiluminescent signal method. Number of participants with ADA to SHP681 in MAD at Day 36 were reported.
Time Frame: Day 36
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Multiple Ascending Dose (MAD): Placebo | Part 2: Multiple Ascending Dose (MAD): 0.2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 0.5 mg/kg | Part 2: Multiple Ascending Dose (MAD): 1 mg/kg | Part 2: Multiple Ascending Dose (MAD): 2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (Q2W)
Number analyzed (Participants) | 12 | 10 | 10 | 8 | 9 | 10 | 9
Participants | 0 | 0 | 1 | 2 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Anti-drug Antibody (ADA) to SHP681 in Multiple Ascending Dose (MAD) at Day 57
Description: Antibody testing was conducted using an electro chemiluminescent signal method. Number of participants with ADA to SHP681 in MAD at Day 57 were reported.
Time Frame: Day 57
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Multiple Ascending Dose (MAD): Placebo | Part 2: Multiple Ascending Dose (MAD): 0.2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 0.5 mg/kg | Part 2: Multiple Ascending Dose (MAD): 1 mg/kg | Part 2: Multiple Ascending Dose (MAD): 2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (Q2W)
Number analyzed (Participants) | 11 | 10 | 10 | 8 | 9 | 10 | 9
Participants | 0 | 0 | 1 | 1 | 1 | 1 | 0

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of SHP681 During Single Ascending Dose (SAD)
Description: Cmax of SHP681 during SAD was reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: Pre-dose, 3, 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672 hours post-dose
Population: Pharmacokinetic (PK) analysis set consisted of participants who received at least 1 dose of SHP681 and had at least 1 evaluable post-dose PK concentration value which was evaluable and interpretable.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter (mcg/mL)
Arm/Group | Part 1: Single Ascending Dose (SAD): 0.2 mg/kg | Part 1: Single Ascending Dose (SAD): 0.5 mg/kg | Part 1: Single Ascending Dose (SAD): 1 mg/kg | Part 1: Single Ascending Dose (SAD): 2 mg/kg | Part 1: Single Ascending Dose (SAD): 4 mg/kg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
Micrograms per milliliter (mcg/mL) | 0.8399 (73.2) | 1.515 (27.7) | 4.200 (26.8) | 8.647 (28.4) | 18.39 (25.2)

7. Secondary Outcome: Time of the Last Measurable Concentration (Tlast) of SHP681 During Single Ascending Dose (SAD)
Description: tlast of SHP681 during SAD was reported.
Time Frame: Pre-dose, 3, 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672 hours post-dose
Population: PK analysis set consisted of participants who received at least 1 dose of SHP681 and had at least 1 evaluable post-dose PK concentration value which was evaluable and interpretable.
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 1: Single Ascending Dose (SAD): 0.2 mg/kg | Part 1: Single Ascending Dose (SAD): 0.5 mg/kg | Part 1: Single Ascending Dose (SAD): 1 mg/kg | Part 1: Single Ascending Dose (SAD): 2 mg/kg | Part 1: Single Ascending Dose (SAD): 4 mg/kg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
Hour | 335.0 [312 to 504] | 504.0 [504 to 672] | 673.0 [671 to 696] | 672.0 [648 to 673] | 672.0 [168 to 673]

8. Secondary Outcome: Time of Maximum Observed Concentration Sampled During a Dosing Interval (Tmax) of SHP681 During Single Ascending Dose (SAD)
Description: tmax of SHP681 during SAD was reported.
Time Frame: Pre-dose, 3, 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672 hours post-dose
Population: as for outcome 7
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 1: Single Ascending Dose (SAD): 0.2 mg/kg | Part 1: Single Ascending Dose (SAD): 0.5 mg/kg | Part 1: Single Ascending Dose (SAD): 1 mg/kg | Part 1: Single Ascending Dose (SAD): 2 mg/kg | Part 1: Single Ascending Dose (SAD): 4 mg/kg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
Hour | 24.00 [24.0 to 96.0] | 72.00 [48.0 to 96.0] | 48.00 [48.0 to 72.0] | 72.00 [48.0 to 96.0] | 72.00 [48.0 to 96.0]

9. Secondary Outcome: Area Under the Curve From the Time of Dosing to the Last Measurable Concentration (AUC0-last) of SHP681 During Single Ascending Dose (SAD)
Description: AUC0-last of SHP681 during SAD was reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: Pre-dose, 3, 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram per milliliter (h*mcg/mL)
Arm/Group | Part 1: Single Ascending Dose (SAD): 0.2 mg/kg | Part 1: Single Ascending Dose (SAD): 0.5 mg/kg | Part 1: Single Ascending Dose (SAD): 1 mg/kg | Part 1: Single Ascending Dose (SAD): 2 mg/kg | Part 1: Single Ascending Dose (SAD): 4 mg/kg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
Hour*microgram per milliliter (h*mcg/mL) | 131.4 (43.7) | 282.1 (31.9) | 794.6 (16.3) | 1722 (25.6) | 3414 (23.5)

10. Secondary Outcome: Area Under the Curve Extrapolated to Infinity (AUC0-inf) of SHP681 During Single Ascending Dose (SAD)
Description: AUC0-inf of SHP681 during SAD was reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: Pre-dose, 3, 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | Part 1: Single Ascending Dose (SAD): 0.2 mg/kg | Part 1: Single Ascending Dose (SAD): 0.5 mg/kg | Part 1: Single Ascending Dose (SAD): 1 mg/kg | Part 1: Single Ascending Dose (SAD): 2 mg/kg | Part 1: Single Ascending Dose (SAD): 4 mg/kg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
h*mcg/mL | 141.0 (36.9) | 288.6 (31.3) | 808.3 (16.4) | 1739 (25.8) | 3446 (23.5)

11. Secondary Outcome: Terminal Half-life (t1/2) of SHP681 During Single Ascending Dose (SAD)
Description: t1/2 of SHP681 during SAD was reported.
Time Frame: Pre-dose, 3, 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672 hours post-dose
Population: as for outcome 7
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 1: Single Ascending Dose (SAD): 0.2 mg/kg | Part 1: Single Ascending Dose (SAD): 0.5 mg/kg | Part 1: Single Ascending Dose (SAD): 1 mg/kg | Part 1: Single Ascending Dose (SAD): 2 mg/kg | Part 1: Single Ascending Dose (SAD): 4 mg/kg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
Hour | 94.50 [64.9 to 109] | 88.40 [76.0 to 104] | 97.10 [90.1 to 124] | 95.40 [87.8 to 116] | 97.80 [86.6 to 127]

12. Secondary Outcome: Average Concentration From Time Zero to 24 Hours Post Dose (Cavg,0-24) of SHP681 During Single Ascending Dose (SAD)
Description: Cavg,0-24 of SHP681 during SAD was reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: Pre-dose, 3, 6, 12, 24 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (mcg/mL)
Arm/Group | Part 1: Single Ascending Dose (SAD): 0.2 mg/kg | Part 1: Single Ascending Dose (SAD): 0.5 mg/kg | Part 1: Single Ascending Dose (SAD): 1 mg/kg | Part 1: Single Ascending Dose (SAD): 2 mg/kg | Part 1: Single Ascending Dose (SAD): 4 mg/kg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
Microgram per milliliter (mcg/mL) | 0.3733 (227.3) | 0.6020 (41.3) | 1.995 (36.0) | 3.193 (43.7) | 7.401 (52.3)

13. Secondary Outcome: First Order Rate Constant Associated With the Terminal (Log-linear) Portion of the Curve (Lambda z) of SHP681 During Single Ascending Dose (SAD)
Description: Lambda z of SHP681 during SAD was reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: Pre-dose, 3, 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: One per hour (1/h)
Arm/Group | Part 1: Single Ascending Dose (SAD): 0.2 mg/kg | Part 1: Single Ascending Dose (SAD): 0.5 mg/kg | Part 1: Single Ascending Dose (SAD): 1 mg/kg | Part 1: Single Ascending Dose (SAD): 2 mg/kg | Part 1: Single Ascending Dose (SAD): 4 mg/kg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
One per hour (1/h) | 0.008156 (23.6) | 0.007907 (14.2) | 0.006945 (12.8) | 0.007050 (10.4) | 0.007011 (15.2)

14. Secondary Outcome: Apparent Total Body Clearance for Extravascular Administration Divided by the Fraction of Dose Absorbed Calculated as Dose Divided by AUC0-inf (CL/F) of SHP681 During Single Ascending Dose (SAD)
Description: CL/F of SHP681 during SAD was reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: Pre-dose, 3, 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Arm/Group | Part 1: Single Ascending Dose (SAD): 0.2 mg/kg | Part 1: Single Ascending Dose (SAD): 0.5 mg/kg | Part 1: Single Ascending Dose (SAD): 1 mg/kg | Part 1: Single Ascending Dose (SAD): 2 mg/kg | Part 1: Single Ascending Dose (SAD): 4 mg/kg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
Liter per hour (L/h) | 0.09810 (22.6) | 0.1188 (42.9) | 0.08856 (20.6) | 0.09909 (33.7) | 0.09689 (25.0)

15. Secondary Outcome: Apparent Volume of Distribution Following Extravascular Administration Divided by the Fraction of Dose Absorbed Calculated as CL/F Divided by Lambda z (Vz/F) of SHP681 During Single Ascending Dose (SAD)
Description: Vz/F of SHP681 during SAD was reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: Pre-dose, 3, 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Part 1: Single Ascending Dose (SAD): 0.2 mg/kg | Part 1: Single Ascending Dose (SAD): 0.5 mg/kg | Part 1: Single Ascending Dose (SAD): 1 mg/kg | Part 1: Single Ascending Dose (SAD): 2 mg/kg | Part 1: Single Ascending Dose (SAD): 4 mg/kg
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
Liter | 12.01 (37.2) | 15.02 (54.7) | 12.75 (27.8) | 14.05 (35.8) | 12.98 (27.2)

16. Secondary Outcome: Average Concentration From Time Zero to 24 Hours Post First Dose (Cavg,0-24) of SHP681 Post First Dose During Multiple Ascending Dose (MAD)
Description: Cavg,0-24 of SHP681 post first dose during MAD was reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: 3, 6, 12, 24 hours post-dose on Day 1
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Part 2: Multiple Ascending Dose (MAD): 0.2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 0.5 mg/kg | Part 2: Multiple Ascending Dose (MAD): 1 mg/kg | Part 2: Multiple Ascending Dose (MAD): 2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (Q2W)
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
mcg/mL | 0.1716 (77.2) | 0.5091 (69.5) | 1.610 (72.0) | 2.108 (39.2) | 4.598 (40.4) | 5.660 (60.7)

17. Secondary Outcome: Observed Concentration at the End of Each Dosing Interval (Immediately Before Next Dose) (Ctrough) of SHP681 for the First 5 Cohorts and Immediately Before 2nd and 3rd Dose of the 6th MAD Cohort During Multiple Ascending Dose (MAD)
Description: Ctrough of SHP681 for the First 5 cohorts and immediately before 2nd and 3rd dose of the 6th MAD cohort during MAD was reported.
Time Frame: Pre-dose on Days 8, 15, 22 and 29
Population: PK analysis set consisted of participants who received at least 1 dose of SHP681 and had at least 1 evaluable post-dose PK concentration value which was evaluable and interpretable. Here the number of participants analyzed signifies participants who were evaluable for this outcome measure at the specific categories.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Part 2: Multiple Ascending Dose (MAD): 0.2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 0.5 mg/kg | Part 2: Multiple Ascending Dose (MAD): 1 mg/kg | Part 2: Multiple Ascending Dose (MAD): 2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (Q2W)
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 9
mcg/mL
  Day 8: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 0
  Day 8 | 0.3523 (39.2) | 0.8432 (28.2) | 1.754 (11.9) | 4.062 (23.5) | 6.949 (20.9) |
  Day 15: number analyzed (Participants) | 10 | 10 | 9 | 9 | 10 | 9
  Day 15 | 0.4688 (27.7) | 1.182 (30.6) | 2.332 (20.6) | 5.312 (14.6) | 9.888 (28.5) | 2.931 (22.9)
  Day 22: number analyzed (Participants) | 10 | 10 | 8 | 9 | 10 | 0
  Day 22 | 0.4593 (26.5) | 1.146 (25.1) | 2.707 (12.3) | 5.249 (18.8) | 13.09 (23.0) |
  Day 29: number analyzed (Participants) | 10 | 10 | 8 | 9 | 10 | 9
  Day 29 | 0.5288 (24.8) | 1.203 (25.8) | 2.659 (14.4) | 5.775 (27.4) | 12.92 (26.7) | 3.109 (22.3)

18. Secondary Outcome: Maximum Concentration During the Dosing Interval Occurring at Tmax (Cmax) of SHP681 Post Fifth Dose During Multiple Ascending Dose (MAD)
Description: Cmax of SHP681 post fifth dose during MAD was reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: 3, 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672 and up to 768 hours post--dose on Day 29
Population: PK analysis set consisted of participants who received at least 1 dose of SHP681 and had at least 1 evaluable post-dose PK concentration value which was evaluable and interpretable. Here the number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Part 2: Multiple Ascending Dose (MAD): 0.2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 0.5 mg/kg | Part 2: Multiple Ascending Dose (MAD): 1 mg/kg | Part 2: Multiple Ascending Dose (MAD): 2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (Q2W)
Number analyzed (Participants) | 10 | 10 | 8 | 9 | 10 | 9
mcg/mL | 0.9710 (38.0) | 2.215 (39.5) | 4.819 (19.6) | 10.38 (34.3) | 24.15 (28.2) | 14.45 (31.5)

19. Secondary Outcome: Time of the Last Measurable Concentration (Tlast) of SHP681 Post Fifth Dose During Multiple Ascending Dose (MAD)
Description: Tlast of SHP681 post fifth dose during MAD was reported.
Time Frame: 3, 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672 and up to 768 hours post--dose on Day 29
Population: as for outcome 18
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 2: Multiple Ascending Dose (MAD): 0.2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 0.5 mg/kg | Part 2: Multiple Ascending Dose (MAD): 1 mg/kg | Part 2: Multiple Ascending Dose (MAD): 2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (Q2W)
Number analyzed (Participants) | 10 | 10 | 8 | 9 | 10 | 9
Hour | 504.0 [504 to 672] | 672.0 [503 to 674] | 672.5 [669 to 674] | 672.0 [672 to 673] | 672.0 [647 to 672] | 672.0 [623 to 768]

20. Secondary Outcome: Time of Maximum Observed Concentration Sampled During a Dosing Interval (Tmax) of SHP681 Post Fifth Dose During Multiple Ascending Dose (MAD)
Description: tmax of SHP681 post fifth dose during MAD was reported.
Time Frame: 3, 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672 and up to 768 hours post--dose on Day 29
Population: as for outcome 18
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 2: Multiple Ascending Dose (MAD): 0.2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 0.5 mg/kg | Part 2: Multiple Ascending Dose (MAD): 1 mg/kg | Part 2: Multiple Ascending Dose (MAD): 2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (Q2W)
Number analyzed (Participants) | 10 | 10 | 8 | 9 | 10 | 9
Hour | 72.00 [12.0 to 168] | 36.00 [3.00 to 96.0] | 48.00 [24.0 to 96.0] | 48.00 [12.0 to 72.0] | 48.00 [48.0 to 72.0] | 72.00 [48.0 to 96.0]

21. Secondary Outcome: Area Under the Curve for the Defined Interval Between Doses (Only Calculated if Interpretable) (AUC0-tau) of SHP681 Post Fifth Dose During Multiple Ascending Dose (MAD)
Description: AUC0-tau of SHP681 post fifth dose during MAD was reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: 3, 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672 and up to 768 hours post--dose on Day 29
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | Part 2: Multiple Ascending Dose (MAD): 0.2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 0.5 mg/kg | Part 2: Multiple Ascending Dose (MAD): 1 mg/kg | Part 2: Multiple Ascending Dose (MAD): 2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (Q2W)
Number analyzed (Participants) | 10 | 10 | 8 | 9 | 10 | 9
h*mcg/mL | 129.6 (33.2) | 282.1 (36.2) | 645.2 (18.7) | 1344 (32.6) | 3297 (24.8) | 2816 (25.9)

22. Secondary Outcome: Area Under the Curve From the Time of Dosing to the Last Measurable Concentration (AUC0-last) of SHP681 Post Fifth Dose During Multiple Ascending Dose (MAD)
Description: AUC0-last of SHP681 post fifth dose during MAD was reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: 3, 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672 and up to 768 hours post--dose on Day 29
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | Part 2: Multiple Ascending Dose (MAD): 0.2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 0.5 mg/kg | Part 2: Multiple Ascending Dose (MAD): 1 mg/kg | Part 2: Multiple Ascending Dose (MAD): 2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (Q2W)
Number analyzed (Participants) | 10 | 10 | 8 | 9 | 10 | 9
h*mcg/mL | 197.8 (29.1) | 435.2 (33.8) | 991.4 (16.3) | 2177 (29.9) | 5456 (22.8) | 3230 (24.7)

23. Secondary Outcome: Area Under the Curve Extrapolated to Infinity (AUC0-inf) of SHP681 Post Fifth Dose During Multiple Ascending Dose (MAD)
Description: AUC0-inf of SHP681 post fifth dose during MAD was reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: 3, 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672 and up to 768 hours post--dose on Day 29
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | Part 2: Multiple Ascending Dose (MAD): 0.2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 0.5 mg/kg | Part 2: Multiple Ascending Dose (MAD): 1 mg/kg | Part 2: Multiple Ascending Dose (MAD): 2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (Q2W)
Number analyzed (Participants) | 10 | 10 | 8 | 9 | 10 | 9
h*mcg/mL | 203.4 (28.5) | 443.1 (33.5) | 1006 (16.3) | 2216 (29.6) | 5548 (22.8) | 3277 (24.5)

24. Secondary Outcome: Average Concentration From Time Zero to 24 Hours Post Dose (Cavg,0-24) of SHP681 During Multiple Ascending Dose (MAD)
Description: Cavg,0-24 of SHP681 during MAD was reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: 3, 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672 and up to 768 hours post--dose on Day 29
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Part 2: Multiple Ascending Dose (MAD): 0.2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 0.5 mg/kg | Part 2: Multiple Ascending Dose (MAD): 1 mg/kg | Part 2: Multiple Ascending Dose (MAD): 2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (Q2W)
Number analyzed (Participants) | 10 | 10 | 8 | 9 | 10 | 9
mcg/mL | 0.6956 (42.3) | 1.683 (36.9) | 3.619 (20.8) | 7.942 (22.3) | 17.04 (23.4) | 7.006 (35.9)

25. Secondary Outcome: Terminal Half-life (t1/2) of SHP681 Post Fifth Dose During Multiple Ascending Dose (MAD)
Description: t1/2 of SHP681 post fifth dose during MAD was reported.
Time Frame: 3, 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672 and up to 768 hours post--dose on Day 29
Population: as for outcome 18
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 2: Multiple Ascending Dose (MAD): 0.2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 0.5 mg/kg | Part 2: Multiple Ascending Dose (MAD): 1 mg/kg | Part 2: Multiple Ascending Dose (MAD): 2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (Q2W)
Number analyzed (Participants) | 10 | 10 | 8 | 9 | 10 | 9
Hour | 96.30 [82.6 to 116] | 108.5 [81.3 to 130] | 103.5 [96.6 to 116] | 105.0 [98.2 to 131] | 106.5 [96.4 to 131] | 99.10 [92.3 to 110]

26. Secondary Outcome: First Order Rate Constant Associated With the Terminal (Log-linear) Portion of the Curve (Lambda z) of SHP681 Post Fifth Dose During Multiple Ascending Dose (MAD)
Description: Lambda z of SHP681 post fifth dose during MAD was reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: 3, 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672 and up to 768 hours post--dose on Day 29
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Part 2: Multiple Ascending Dose (MAD): 0.2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 0.5 mg/kg | Part 2: Multiple Ascending Dose (MAD): 1 mg/kg | Part 2: Multiple Ascending Dose (MAD): 2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (Q2W)
Number analyzed (Participants) | 10 | 10 | 8 | 9 | 10 | 9
1/h | 0.007215 (9.4) | 0.006667 (14.3) | 0.006633 (6.3) | 0.006416 (8.7) | 0.006473 (9.8) | 0.006922 (5.5)

27. Secondary Outcome: Apparent Total Body Clearance Following Extravascular Administration Divided by the Fraction of Dose Absorbed Calculated as Dose Divided by AUCtau (CL/F) of SHP681 Post Fifth Dose During Multiple Ascending Dose (MAD)
Description: CL/F of SHP681 post fifth dose during MAD was reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: 3, 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672 and up to 768 hours post--dose on Day 29
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Part 2: Multiple Ascending Dose (MAD): 0.2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 0.5 mg/kg | Part 2: Multiple Ascending Dose (MAD): 1 mg/kg | Part 2: Multiple Ascending Dose (MAD): 2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (Q2W)
Number analyzed (Participants) | 10 | 10 | 8 | 9 | 10 | 9
L/h | 0.1225 (38.5) | 0.1366 (53.5) | 0.1141 (21.3) | 0.1226 (35.5) | 0.09547 (27.3) | 0.1100 (19.6)

28. Secondary Outcome: Apparent Volume of Distribution Following Extravascular Administration Divided by the Fraction of Dose Absorbed Calculated as CL/F Divided by Lambda z (Vz/F) of SHP681 Post Fifth Dose During Multiple Ascending Dose (MAD)
Description: Vz/F of SHP681 post fifth dose during MAD was reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: 3, 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672 and up to 768 hours post--dose on Day 29
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Part 2: Multiple Ascending Dose (MAD): 0.2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 0.5 mg/kg | Part 2: Multiple Ascending Dose (MAD): 1 mg/kg | Part 2: Multiple Ascending Dose (MAD): 2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (Q2W)
Number analyzed (Participants) | 10 | 10 | 8 | 9 | 10 | 9
Liter | 16.99 (39.4) | 20.48 (56.4) | 17.21 (24.0) | 19.12 (42.2) | 14.75 (30.8) | 15.89 (17.8)

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to follow-up (Day 29 for SAD / Day 57 for MAD)
Arm/Group | Part 1: Single Ascending Dose (SAD): Placebo | Part 1: Single Ascending Dose (SAD): 0.2 mg/kg | Part 1: Single Ascending Dose (SAD): 0.5 mg/kg | Part 1: Single Ascending Dose (SAD): 1 mg/kg | Part 1: Single Ascending Dose (SAD): 2 mg/kg | Part 1: Single Ascending Dose (SAD): 4 mg/kg | Part 2: Multiple Ascending Dose (MAD): Placebo | Part 2: Multiple Ascending Dose (MAD): 0.2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 0.5 mg/kg | Part 2: Multiple Ascending Dose (MAD): 1 mg/kg | Part 2: Multiple Ascending Dose (MAD): 2 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (Q2W)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/12 | 0/10 | 0/10 | 0/10 | 0/10 | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/12 | 0/10 | 0/10 | 0/10 | 1/10 | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 3/5 | 3/5 | 2/5 | 4/5 | 3/5 | 2/5 | 9/12 | 8/10 | 3/10 | 6/10 | 5/10 | 9/12 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Single Ascending Dose (SAD): Placebo (N=5) | Part 1: Single Ascending Dose (SAD): 0.2 mg/kg (N=5) | Part 1: Single Ascending Dose (SAD): 0.5 mg/kg (N=5) | Part 1: Single Ascending Dose (SAD): 1 mg/kg (N=5) | Part 1: Single Ascending Dose (SAD): 2 mg/kg (N=5) | Part 1: Single Ascending Dose (SAD): 4 mg/kg (N=5) | Part 2: Multiple Ascending Dose (MAD): Placebo (N=12) | Part 2: Multiple Ascending Dose (MAD): 0.2 mg/kg (N=10) | Part 2: Multiple Ascending Dose (MAD): 0.5 mg/kg (N=10) | Part 2: Multiple Ascending Dose (MAD): 1 mg/kg (N=10) | Part 2: Multiple Ascending Dose (MAD): 2 mg/kg (N=10) | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (N=12) | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (Q2W) (N=10)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Single Ascending Dose (SAD): Placebo (N=5) | Part 1: Single Ascending Dose (SAD): 0.2 mg/kg (N=5) | Part 1: Single Ascending Dose (SAD): 0.5 mg/kg (N=5) | Part 1: Single Ascending Dose (SAD): 1 mg/kg (N=5) | Part 1: Single Ascending Dose (SAD): 2 mg/kg (N=5) | Part 1: Single Ascending Dose (SAD): 4 mg/kg (N=5) | Part 2: Multiple Ascending Dose (MAD): Placebo (N=12) | Part 2: Multiple Ascending Dose (MAD): 0.2 mg/kg (N=10) | Part 2: Multiple Ascending Dose (MAD): 0.5 mg/kg (N=10) | Part 2: Multiple Ascending Dose (MAD): 1 mg/kg (N=10) | Part 2: Multiple Ascending Dose (MAD): 2 mg/kg (N=10) | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (N=12) | Part 2: Multiple Ascending Dose (MAD): 4 mg/kg (Q2W) (N=10)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 4 (8) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (6) | 0 (0)
Application site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 3 (4) | 2 (2) | 1 (1) | 3 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 1 (2) | 1 (2) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT03859323/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/23/NCT03859323/SAP_001.pdf